CLINICAL TRIAL: NCT03974503
Title: Characterization of Sleep With Trauma Nightmares Using Ambulatory Sleep Measurement
Brief Title: Understanding Trauma Nightmares Using In-Home Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-018-18F; IK2CX001874 (NIH)
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Nightmares; Stress Disorders, Post-Traumatic; Actigraphy; Respiratory Sinus Arrhythmia; Veterans
Keywords: Nightmares; Cognitive Behavioral Therapy; PTSD; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Arrhythmia, Sinus | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two cognitive-behavioral treatments for sleep and nightmares.
Who Masked: Outcomes Assessor
Masking Description: Assessors at the post-treatment and follow-up assessment will not be aware of what treatment the participants received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exposure, Relaxation, and Rescripting Therapy (ERRT) (Experimental): Exposure, Relaxation, & Rescripting Therapy (ERRT) will be conducted once a week for five consecutive weeks for approximately one hour per session. Each treatment session focuses on one of the following topics/skills: psycho-education and investment in treatment, sleep behavior modification, Progressive Muscle Relaxation, diaphragmatic breathing, exposure to the trauma-nightmare, rescription, and treatment maintenance planning.
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy
- Sleep and Nightmare Management (Active Comparator): This treatment protocol has amounts of therapist contact, handouts, and homework between sessions equivalent to those in ERRT. The protocol contains psychoeducation about sleep disturbances and trauma-related nightmares, including their distressing nature, chronicity, and impact on sleep and daytime functioning. Additionally, basic sleep behavior modification are presented. No nightmare content or rescripting will be explicitly discussed, and the diaphragmatic breathing techniques will be omitted from this protocol.
  Interventions: Behavioral: Sleep and Nightmare Management

INTERVENTIONS:
Behavioral: Exposure, Relaxation, and Rescripting Therapy — ERRT is a weekly 5-session treatment aimed at reducing chronic trauma nightmares and sleep disturbances in trauma-exposed adults.
  Other Names: ERRT
  Arms: Exposure, Relaxation, and Rescripting Therapy (ERRT)
Behavioral: Sleep and Nightmare Management — This is a manualized protocol developed to be of similar length but exclude the active components of standard ERRT.
  Arms: Sleep and Nightmare Management

SUMMARY:
Trauma-related nightmares in Veterans are associated with poor clinical outcomes, greater substance use, and increased risk of suicide. In spite of an urgent need to reduce the burden of trauma-related nightmares, the underlying physiological changes associated with them are poorly understood, and there are no clear evidence-based recommendations for their treatment. Limitations of current assessment procedures represent a barrier to improved care. In-laboratory sleep studies rarely capture nightmares, limiting the knowledge about them and their response to treatment. This study addresses these limitations by using extended, in-home sleep monitoring to capture sleep data associated with nightmare reports in Veterans, and assessing how these features are altered throughout a cognitive-behavioral nightmare treatment. Results from this study will increase understanding of trauma-related nightmares, and advance strategies for personalizing symptom management for Veterans.

DETAILED DESCRIPTION:
There is a critical need for continued research to better understand trauma-related nightmares with the goal of developing personalized treatment plans. Limitations of current assessment procedures present a significant barrier to improved care. In-laboratory sleep studies rarely capture nightmares and cannot assess change over time, reducing the knowledge of phenotypic markers of nightmares to guide treatment. Therefore, there is a need to assess sleep over multiple nights in the home environment, where nightmares occur. This study aims to significantly enrich knowledge about trauma-related nightmares by using a zero-burden, multi-night, objective sleep measurement method within Veterans' usual sleeping environment prior to and during an evidence-based cognitive-behavioral intervention for nightmares. This study has two primary aims: 1) to identify, with greater precision than previously possible, objective features of sleep associated with trauma-related nightmare occurrences; and 2) to use the treatment for nightmares as interventional probes to determine whether and how changes in sleep physiological parameters identified in Aim 1 covary with changes in subjective nightmare frequency and severity.

The study will include 80 trauma-exposed Veterans reporting with trauma-related nightmares. Eligible participants will monitor their sleep for a week using a multi-night mattress actigraphy implemented in their home. Mattress actigraphy, which measures movements using accelerometers embedded in a mattress topper, employs no body surface sensors. Therefore, this system represents a truly zero-burden method for obtaining intensive longitudinal sleep measurement. During the week of sleep monitoring, participants also will complete one-night of polysomnography (PSG) sleep assessment to calibrate the actigraphic sleep efficiency and to identify untreated sleep apnea. These methods will be used to investigate candidate physiological parameters associated with trauma-related nightmares. After establishing the levels of these candidate markers, this project will assess the impact of a cognitive-behavioral treatment, Exposure, Relaxation, and Rescripting Therapy (ERRT), on the subset of markers which can be measured continuously over the course of the treatment. Participants will be randomized to five weeks of active treatment (ERRT; n = 40) or to five weeks of the comparison treatment (sleep and nightmare management; n = 40). Throughout the course of treatment, participants will continue to sleep while monitored by the mattress actigraphy system. Upon completion of treatment, a post-treatment and follow-up assessment will assess subjective symptom change. Results from this study will provide important information to facilitate increased understanding of the phenomenology, pathophysiology, and treatment of nightmares in trauma-exposed Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Be a Veteran enrolled to receive VA medical care at the Minneapolis VA Health Care System
* Have stable housing for the duration of the study period
* Have experienced any traumatic event meeting Criterion A for PTSD at least three months before the baseline assessment
* Meet criteria for a current PTSD diagnosis or subthreshold PTSD diagnosis
* Self-report experiencing trauma-related nightmares at least once per week for the past month, that are mostly-remembered and that cause awakening
* Self-report global sleep disturbance indicated by a score of 5 or greater on the Pittsburgh Sleep Quality Index (PSQI)
* Be stable on any psychoactive medications for a minimum of two weeks before the baseline assessment

Exclusion Criteria:

* Inability to provide fully-informed written consent to participate and/or a bed partner does not agree to mattress recording during the in-home portion of the study
* Medical conditions that limit ability to apply the treatment e.g., needing a health aide or caregiver to record sleep diaries, unable to get out of bed without assistance
* Current pregnancy and/or birth of a child within the previous 6 months
* Current alcohol or illicit substance use disorders or early remission (at least 3 months abstinent)
* Active suicidal or homicidal ideation
* A history of any bipolar disorder spectrum disorder or psychotic disorder
* Hospitalization for a mental health disorder in the past 2 months
* Enrolled in current PTSD-focused treatment (e.g., Cognitive Processing Therapy or Prolonged Exposure), current nightmare treatment or a history of treatment failure with a cognitive-behavioral nightmare intervention
* Veterans may also be excluded from participation if they have been identified by the local VA disruptive behavior committee to have displayed disruptive, threatening and/or violent behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Change in Actigraphy-derived sleep efficiency (SE) | Nightly up to 7 weeks (Baseline through 1-week post treatment assessment)
  Mattress actigraphy will be continuously recorded during the study period. Sleep efficiency is defined as the ratio of the aggregate duration of quiescent sleep periods divided by the duration of the total in bed period. Lower sleep efficiency indicates worse sleep.
Change in Actigraphy-derived respiratory sinus arrhythmia (RSA) | Nightly (Baseline until 1-week post treatment assessment; 7 weeks)
  Mattress actigraphy will be continuously recorded during the study period. RSA is the high frequency powers of heart period variability (0.15-0.4 Hz). Lower RSA indicates more cardiac vagal withdrawal.
Change in Nightmare Frequency | Baseline past week; Nightly during baseline; 1-week post-treatment; 3-month follow-up treatment period
  This fill-in-the-blank variable assesses the number of nightmares experienced in the past week (range = 0 - X nightmares) at each assessment (baseline, one week following treatment, and three months following treatment). Nightly reports will be collected from daily sleep diaries and pushes to event markers during the night.

SECONDARY OUTCOMES:
Change in PTSD Symptom Severity | Baseline, 1-week post-treatment, 3-month follow-up
  Change in PTSD Symptoms will be assessed using the Clinician-Administered PTSD Scale DSM 5 (CAPS-5) and the self-report PTSD Symptom Checklist. The items on the CAPS-5 are on a 5-point scale (0 - 4), (possible range: 0-80). A symptom is considered present if the severity is rated 2 or higher. Total scores are comprised of four factors (reexperiencing, avoidance, cognitive/emotional and hyperarousal)
Change in Nightmare Severity | Baseline; Nightly during baseline; 1-week post-treatment; 3-month follow-up treatment period
  The variable from the Trauma-Related Nightmare Survey assesses the severity of the nightmares experienced in the past week (range = 0 - 4) at each assessment (baseline, one week following treatment, and three months following treatment). Nightly reports of nightmare severity will be collected from daily sleep diaries. Higher scores indicate greater nightmare-related severity.

OTHER OUTCOMES:
Home-based overnight polysomnography | Baseline
  Nox A1 portable polysomnography system (Nox Medical, Reykjavik, Iceland) used to record sleep stage measures and patterns of arousals, to calibrate sleep efficiency derived from the mattress system, and to detect sleep apnea.
Change in Global Sleep Quality | Baseline, 1-week post-treatment, 3-month follow-up
  Change in sleep Quality will be assessed using the Pittsburgh Sleep Quality Index, a 19-item self-report measure assessing qualities and problems associated with sleep in the past month. A global sleep quality score is obtained by summing seven component scores. Higher scores reflect poorer sleep quality. The global score ranges from 0 to 21, with a cut-off score of 5 as distinguishing "good" sleepers from "poor" sleepers.
  The addendum is used in conjunction with the PSQI for use with trauma-exposed participants and assesses the presence of seven trauma-related sleep disturbances.
Change in self-report depression symptoms | Baseline, 1-week post-treatment, 3-month follow-up
  The patient health questionnaire (PHQ-9), is a 9-item self-report instrument used to assess depression severity. Items are scored 0 to 3, with the total score being the sum of the 9 items. Higher scores indicate greater depression severity, with a score of 10 or greater considered major depression, and scores of 20 or more is severe major depression.
Change in Nightmare Effects | Baseline, 1-week post-treatment, 3-month follow-up
  Change in the impact of nightmares will be assessed using the change in Nightmare Effects Survey, an 11 item Likert-type questionnaire designed to assess the impact of nightmares on 11 areas of life including work, social, and leisure activities. Total scores range from 0 to 44, with higher scores indicating greater level of nightmare-related impairment.
Change in Fear of Sleep | Baseline, 1-week post-treatment, 3-month follow-up
  Change in fear of sleep will be assessed using the Fear of Sleep Inventory, a 23-item self-report measure that assesses trauma-related thoughts and activities associated with sleep and the occurrence of traumas associated with the bedroom or sleep. Total scores range from 0 to 92, with higher scores indicating greater fear of sleep.
Change in suicidal ideation | Baseline, 1-week post-treatment, 3-month follow-up
  Change in suicidal ideation will be assessed using the Depressive Symptom Index: Suicidality Subscale (DSI-SS). The four items of the DSI-SS are scored on a 0-3 scale, with total possible sum scores ranging from 0-12; higher scores indicate greater severity of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Elizabeth Miller, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhn E, Miller KE, Puran D, Wielgosz J, YorkWilliams SL, Owen JE, Jaworski BK, Hallenbeck HW, McCaslin SE, Taylor KL. A Pilot Randomized Controlled Trial of the Insomnia Coach Mobile App to Assess Its Feasibility, Acceptability, and Potential Efficacy. Behav Ther. 2022 May;53(3):440-457. doi: 10.1016/j.beth.2021.11.003. Epub 2021 Nov 19. PMID 35473648
- [Background] Tighe CA, Berlin GS, Boland EM, Miller KE, Bramoweth AD. Identifying predictors of the amount of veteran participation in cognitive behavioral therapy for insomnia in the Veterans Affairs health care system. Psychol Serv. 2024 Aug;21(3):581-588. doi: 10.1037/ser0000818. Epub 2023 Nov 2. PMID 37917476
- [Background] Miller KE, So CJ, Brownlow JA, Woodward SH, Gehrman PR. Neighborhood disadvantage is associated with sleep disturbance in a sample of trauma-exposed Veterans. Sleep Health. 2023 Oct;9(5):634-637. doi: 10.1016/j.sleh.2023.06.006. Epub 2023 Jul 31. PMID 37532605
- [Background] Miller KE, Bolstad CJ, Carlile JA, Balliett NE, Trivedi S, Davis JL, Schubert J, Krieg C, Shah M. Providers' use and perceived benefits and barriers of delivering cognitive behavioral therapy for nightmares (CBT-N) to veterans. Psychol Serv. 2025 Sep 15:10.1037/ser0000994. doi: 10.1037/ser0000994. Online ahead of print. PMID 40952699
- [Background] So CJ, Bolstad CJ, Miller KE. Status of Imagery Rehearsal Therapy and Other Interventions for Nightmare Treatment in PTSD. Curr Psychiatry Rep. 2025 Nov;27(11):671-678. doi: 10.1007/s11920-025-01639-z. Epub 2025 Sep 11. PMID 40932590
- [Background] Miller KE, Boland EM, Barilla H, Ross RJ, Kling MA, Bhatnagar S, Gehrman PR. Ecological momentary assessment of daily affect, stress, and nightmare reports among combat-exposed Veterans. Dreaming. 2024;34(4):307-317. doi: 10.1037/drm0000281. PMID 39950038
- [Background] So CJ, Miller KE, Gehrman PR. Sleep Disturbances Associated With Posttraumatic Stress Disorder. Psychiatr Ann. 2023 Nov 1;53(11):491-495. doi: 10.3928/00485713-20231012-01. PMID 38293647
- [Background] Miller KE, Tamayo G, Arsenault N, Jamison AL, Woodward SH. Longitudinal profiles of sleep during residential PTSD treatment. Sleep Med. 2023 Jun;106:52-58. doi: 10.1016/j.sleep.2023.03.020. Epub 2023 Mar 31. PMID 37044001
- [Background] Brownlow JA, Miller KE, Ross RJ, Barilla H, Kling MA, Bhatnagar S, Mellman TA, Gehrman PR. The association of polysomnographic sleep on posttraumatic stress disorder symptom clusters in trauma-exposed civilians and veterans. Sleep Adv. 2022 Aug 11;3(1):zpac024. doi: 10.1093/sleepadvances/zpac024. eCollection 2022. PMID 36171859
- [Background] Brownlow JA, Klingaman EA, Miller KE, Gehrman PR. Trauma type as a risk factor for insomnia in a military population. J Affect Disord. 2022 Jul 1;308:65-70. doi: 10.1016/j.jad.2022.04.018. Epub 2022 Apr 9. PMID 35413357
- [Background] Miller KE, Ross RJ, Harb GC. Lucid Dreams in Veterans With Posttraumatic Stress Disorder Include Nightmares. Dreaming. 2021 Jun;31(2):117-127. PMID 37363340
- [Background] Polyne NC, Miller KE, Brownlow J, Gehrman PR. Insomnia: Sex differences and age of onset in active duty Army soldiers. Sleep Health. 2021 Aug;7(4):504-507. doi: 10.1016/j.sleh.2021.03.003. Epub 2021 Apr 15. PMID 33867309
- [Background] Brownlow JA, Miller KE, Gehrman PR. Treatment of Sleep Comorbidities in Posttraumatic Stress Disorder. Curr Treat Options Psychiatry. 2020 Sep;7(3):301-316. doi: 10.1007/s40501-020-00222-y. Epub 2020 Jun 12. PMID 33552844
- [Background] Miller KE, Babler L, Maillart T, Faerman A, Woodward SH. Sleep/Wake Detection by Behavioral Response to Haptic Stimuli. J Clin Sleep Med. 2019 Nov 15;15(11):1675-1681. doi: 10.5664/jcsm.8038. PMID 31739859
- [Background] Miller KE, Brownlow JA, Gehrman PR. Sleep in PTSD: treatment approaches and outcomes. Curr Opin Psychol. 2020 Aug;34:12-17. doi: 10.1016/j.copsyc.2019.08.017. Epub 2019 Aug 23. PMID 31541965

DOCUMENTS (1):
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03974503/ICF_000.pdf